CLINICAL TRIAL: NCT00002017
Title: Immunomodulation of HIV-1 Infected Individuals With PEG-Interleukin-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 072A; COH-010-0790
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-08

CONDITIONS: HIV Infections
Keywords: Polyethylene Glycols; Interleukin-2
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2, Polyethylene Glycolated

SUMMARY:
To evaluate the safety and immunological effects of polyethylene glycolated-interleukin-2 (PEG-IL-2) on asymptomatic (without symptoms) HIV-seropositive patients who are taking zidovudine (AZT). To enhance measures of immune function with well-tolerated doses of PEG-IL-2, an immunomodulator, in a regimen designed to allow its use in outpatients with normal daily activity (i.e., full-time employment, etc.). Recombinant IL-2 (without PEG modification) was administered to HIV-infected patients by daily intradermal injection. At the low doses used, this was non-toxic, well-tolerated, and gave a systemic response as measured by natural killer cell and lymphokine-activated killer cell activity, but required daily administration. In the current study, the PEG modification of IL-2 is used since it has a much longer prolonged half-life compared with the non-PEG compound, without loss of functional activity.

DETAILED DESCRIPTION:
Recombinant IL-2 (without PEG modification) was administered to HIV-infected patients by daily intradermal injection. At the low doses used, this was non-toxic, well-tolerated, and gave a systemic response as measured by natural killer cell and lymphokine-activated killer cell activity, but required daily administration. In the current study, the PEG modification of IL-2 is used since it has a much longer prolonged half-life compared with the non-PEG compound, without loss of functional activity.

In the first, dose-escalation phase of the study, PEG-IL-2 is injected into the skin of the back by either the intradermal (ID) or subcutaneous (SC) route, to establish an optimal dose (which when given ID results in local induration = or > 25 mm without significant toxicity). The ID and SC routes are compared for systemic effect and toxicity. In the second phase of the study, the PEG-IL-2 is administered for 6-8 weeks using the optimal dosage, frequency, and route determined in the initial phase (probably 2-3 times per week) while local and systemic effects are monitored. These include measures of viral titer, peripheral blood mononuclear cell phenotype, CBC and CD4 counts, and in vitro cytotoxicity assays.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* Necessary topical agents such as nystatin, clotrimazole, and acyclovir.
* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Oral antibiotics for PCP prophylaxis if hematologically stable for = or > 30 days prior to study entry.
* Necessary systemic agents for the treatment of other chronic disorders, such as diabetes or asthma.

Patients must have:

* HIV-1 seropositivity.
* Asymptomatic.
* No opportunistic infection for 8 weeks prior to study entry.
* Been on azidothymidine (AZT) (= or > 500 mg/day) for at least 8 weeks prior to beginning interleukin-2 (IL-2), with stable CD4 cell counts.

Prior Medication:

Allowed:

* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active, life-threatening opportunistic infection (OI) with bacterial, viral, fungal, or protozoan pathogens.
* Fever = or > 101 F. within 10 days prior to study entry.
* Significant central nervous system (CNS) disease including AIDS dementia, psychiatric disability, or seizure disorder.
* Significant cardiac disease (New York Heart Association Stage III or IV).
* Significant pulmonary disease (Forced Expiratory Volume < 75 percent.
* Weight loss = or > 10 percent within last 3 months.

Concurrent Medication:

Excluded:

* Systemic therapy for opportunistic infection (OI).

Patients with the following are excluded:

* Presence of antibody to interleukin-2 (IL-2).
* Diseases or symptoms listed in Exclusion Co-Existing Conditions.

Prior Medication:

Excluded within 12 weeks prior to study entry:

* Other immunomodulators.
* Corticosteroids.
* Other experimental therapy.
* Anti-neoplastic chemotherapy.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Rockefeller Univ, New York, New York, United States

REFERENCES:
- [Background] Teppler H, Montana A, Meyn P, Kaplan G, Cohn ZA. Prolonged immunostimulatory effect of low dose PEG interleukin-2 in HIV-infected individuals. Int Conf AIDS. 1992 Jul 19-24;8(2):B162 (abstract no PoB 3453)
- [Derived] Zhang W, Ruan J, Zhang R, Zhang M, Hu X, Han Z, Ruan Q. Association between age-related hearing loss with tinnitus and cognitive performance in older community-dwelling Chinese adults. Psychogeriatrics. 2022 Nov;22(6):822-832. doi: 10.1111/psyg.12889. Epub 2022 Sep 8. PMID 36075585
- [Derived] Zhang W, Ruan J, Zhang R, Zhang M, Hu X, Yu Z, Han Z, Ruan Q. Age-Related Hearing Loss With Tinnitus and Physical Frailty Influence the Overall and Domain-Specific Quality of Life of Chinese Community-Dwelling Older Adults. Front Med (Lausanne). 2021 Oct 21;8:762556. doi: 10.3389/fmed.2021.762556. eCollection 2021. PMID 34746196
- [Derived] Ruan Q, Chen J, Zhang R, Zhang W, Ruan J, Zhang M, Han C, Yu Z. Heterogeneous Influence of Frailty Phenotypes in Age-Related Hearing Loss and Tinnitus in Chinese Older Adults: An Explorative Study. Front Psychol. 2021 Feb 16;11:617610. doi: 10.3389/fpsyg.2020.617610. eCollection 2020. PMID 33664689